CLINICAL TRIAL: NCT04931407
Title: A Feasibility Study in Chronically Fatigued Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Diakonhjemmet Hospital (Other); Norwegian School of Sport Sciences (Other); Norwegian University of Science and Technology (Other); University of Alberta (Other); UiT The Arctic University of Norway (Other)
Responsible Party: Principal Investigator, Lene Thorsen, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 153665
Record Dates: First submitted 2021-04-16; First posted 2021-06-18 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Fatigue; Lymphoma
Keywords: exercise; chronic fatigue; lymphoma; cancer survivors; nutrition; cognitive therapy; patient education
MeSH Terms: conditions — Fatigue; Lymphoma; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interdisciplinary complex intervention (Experimental): The intervention includes patient education, physical exercise, a group-based cognitive behavioral program and individual nutritional counseling
  Interventions: Other: A 12-week interdisciplinary complex intervention

INTERVENTIONS:
Other: A 12-week interdisciplinary complex intervention — The intervention will last for 12 weeks and includes four components; patient education, physical exercise, cognitive behavioral program and nutritional counseling.
  The patient education will include an online 2-hours group-based patient-education sessions in week 1.
  The physical exercise program includes two weekly exercise sessions, one supervised by a physiotherapist and one unsupervised, including aerobic exercise, resistance exercise and psychometric physiotherapy. Half of the intervention group (N=7) will perform the supervised exercise session individually with a physiotherapist in the municipality, while the other half (n=8) will exercise in online groups lead by physiotherapists.
  The cognitive behavioral program will begin in week 3 and include six group-based online sessions every week lead by a clinical psychologist.
  The nutritional counseling will include three individual digital nutrition counselling sessions in week 2, 6 and 10 by a clinical dietitian.

SUMMARY:
Improved cancer survival has led to increased attention on long-term health and quality of life (QoL) among the survivors. Both the cancer diagnosis and intensive treatments increase the risk of late effects which may interfere with daily physical, psychological and social functioning, and thereby negatively affect their QoL. Well-documented late-effects among cancer survivors are second cancer, cardio-vascular disease, pain, hormone disturbances, mental distress and chronic fatigue (CF).

CF is a subjective experience of substantial lack of energy, exhaustion and cognitive difficulties lasting for six months or longer. CF is one of the most common and distressing late effects after cancer, affecting 15-35 % of survivors, often for years beyond treatment. Despite the high prevalence and the huge negative consequences of CF on daily functioning and QoL and the economic and societal costs, effective treatment of CF and standardized follow-up care are currently lacking.

CF is a complex condition best understood as a multifactorial phenomenon. Our and other research groups have examined various cohorts of cancer survivors in order to identify behavioral-, psychological-, and biological factors associated with CF, that can form the basis for targeted interventions. So far, few treatable biological factors have been identified, even though immune activation, flattened diurnal cortisol slopes and a blunted cortisol response to stress have been demonstrated in small studies among cancer survivors suffering from CF. On the other hand, several modifiable behavioral factors including emotional distress, physical inactivity, sleep disturbances and unhealthy diets are found to be associated with CF. So far, most of the interventions aiming to reduce fatigue during and shortly after cancer treatment have targeted only one of these factors at a time, with small to moderate effect sizes. No prior study has examined if CF in cancer survivors is better treated by a complex intervention targeting combinations of these factors, an approach which seems logical due to the complexity of the symptom.

The Division of Cancer Medicine at Oslo University Hospital (OUH) presently offers limited rehabilitation programs, including patient education, physical exercise, cognitive behavioral program and nutrition counselling to cancer survivors with CF. However, these programs are not offered as an interdisciplinary intervention integrated in a standardized patient care pathway, and the effects of these interventions have not been assessed. Based on the investigators clinical experience and published studies on single-targeted interventions, the investigators hypothesize that a complex intervention including psycho-educational elements, physical exercise and nutrition counseling delivered as a standardized patient care pathway is well-founded and doable, and will improve fatigue, functioning and QoL in cancer survivors with CF.

During the fall of 2021, the investigators will conduct a randomized controlled trial (RCT) with the overall objective to improve fatigue in lymphoma survivors with CF. To uncover strengths and weaknesses with the planned RCT, i.e. the inclusion procedures, the assessments and the complex intervention, the investigators are now conducting a small one-armed feasibility study before the RCT during spring 2021.

ELIGIBILITY:
Seven lymphoma survivors will be included, with the same inclusion criteria as in the planned RCT:

Inclusion Criteria:

* Survivors of Hodgkin and aggressive non-Hodgkin lymphoma, diagnosed 2014 or 2019 (n=7)
* 18-65 years at diagnosis, and 19-67 years at participation.
* CF measured by Chalder FQ.
* Curatively treated, more than 2 years since last treatment.
* Participation approval from oncologist.

Exclusion Criteria:

* Indolent non-Hodgkin lymphoma.
* Fatigue more than one year before the cancer diagnosis.
* Ongoing cancer treatment, relapse or second cancer, somatic/physical conditions (i.e. severe heart failure/disease, lung disease, use of wheelchair /crutches).
* Psychiatric disorders (i.e. severe depression, schizophrenia), substance abuse disorder.

In addition, eight cancer survivors with various diagnosis, will be included from a waiting list for rehabilitation at the Cancer Rehabilitation Centre at Aker hospital.

Ages: 19 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | The week before the intervention period (week 0)
  Assessed by the number who consent to participate
Inclusion rate | The week before the intervention period (week 0)
  Assessed by the number of consenting participants who are included (i.e. have chronic fatigue according to the Fatigue Questionnaire, and are cleared for participation by oncologist after the medical screening).
Completion rate | The week before the intervention period (week 0)
  Assessed by the number of consenting participants consenting patients who complete any measurement at the final assessment
Strengths and weaknesses with the inclusion procedure: participants | Week 4
  Assessed by structured conversations with the participants
Strengths and weaknesses with the inclusion procedure: study personnel | Week 4
  Assessed by structured conversations with the study personnel
Feasibility of the patient education session: participants | Week 4
  Strengths, weaknesses, and usefulness of the contents in the education session will be assessed by structured conversations with the participants after the patient education session.
Feasibility of the patient education session: presenters | Week 4
  Strengths, weaknesses, and usefulness of the contents in the education session will be assessed by structured conversations with the presenters after the patient education session.
Feasibility of the exercise program part one (week 1-3): participants | Week 4
  Strengths and weaknesses with the exercise program will be evaluated through structured conversations with the participants
Feasibility of the exercise program part one (week 1-3): physiotherapists | Week 4
  Strengths and weaknesses with the exercise program will be evaluated through structured conversations with the physiotherapists
Feasibility of the exercise program part two (week 4-7): participants | Week 8
  Strengths and weaknesses with the exercise program will be evaluated through structured conversations with the participants
Feasibility of the exercise program part two (week 4-7): physiotherapists | Week 8
  Strengths and weaknesses with the exercise program will be evaluated through structured conversations with the physiotherapists
Compliance to the cognitive behavioral therapy groups sessions | Week 8
  Participation to the cognitive behavioral therapy groups sessions will be registered by the study coordinators/psychologists..
Feasibility of the cognitive behavioral therapy groups sessions: participants | Week 8
  Strengths, weaknesses, and usefulness of the groups sessions will be assessed by structured conversations with the participants after the last group session
Feasibility of the cognitive behavioral therapy groups sessions: psychologists | Week 8
  Strengths, weaknesses, and usefulness of the groups sessions will be assessed by structured conversations with the psychologists after the last group session
Compliance to the nutrition counseling | Week 11
  Participation rate of the individual nutrition counseling sessions will be registered by the clinical dietitian.
Feasibility of the nutrition counseling: participants | Week 11
  Strengths, weaknesses, and usefulness of the contents in the sessions will be assessed by structured conversations with the participants after the last counseling session.
Feasibility of the nutrition counseling: clinical dietitian | Week 11
  Strengths, weaknesses, and usefulness of the contents in the sessions will be assessed by structured conversations with the clinical dietitian after the last counseling session.
Compliance to the exercise program: attendance | Week 13
  Registered by the physiotherapists in an exercise log
Compliance to the exercise program: intensity during the aerobic exercise intervals | Week 13
  Registered by pulse sensors
Compliance to the exercise program: implementation of the strength training exercises | Week 13
  Registered by the physiotherapists in an exercise log
Feasibility of the exercise program part three (week 8-12): participants | Week 13
  Strengths and weaknesses with the exercise program will be evaluated through structured conversations with the participants
Feasibility of the exercise program part three (week 8-12): physiotherapists | Week 13
  Strengths and weaknesses with the exercise program will be evaluated through structured conversations with the physiotherapists
Feasibility of the questionnaires | Week 13
  Strengths and weaknesses with the questionnaire will be evaluated through structured conversations with the participants.
Feasibility of the physical tests: participants | Week 13
  Strengths and weaknesses with the tests will be evaluated through structured conversations with the participants.
Feasibility of the physical tests: physiotherapists | Week 13
  Strengths and weaknesses with the tests will be evaluated through structured conversations with the physiotherapists conducting the tests.
Compliance to the physical tests | Week 13
  Assessed by the completion rate of the physical tests (i.e. the number of participants who conduct the tests as planned).
Completeness of the questionnaires | Week 13
  Assessed by the completion rate of the questionnaire (i.e. proportion of missing).

SECONDARY OUTCOMES:
Change in level of fatigue | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by Chalder Fatigue Questionnaire. Total score range from 0 to 33, with increasing score implying more fatigue.
Change in level of fatigue | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by Chalder Fatigue Questionnaire. Total score range from 0 to 33, with increasing score implying more fatigue.
Change in level of fatigue | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by Chalder Fatigue Questionnaire. Total score range from 0 to 33, with increasing score implying more fatigue.
Change in daily functioning and global quality of life | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30). Scores range fro 0 to 100, a higher score represents a higher (better) level of functioning or a higher (worse) level of symptoms.
Change in daily functioning and global quality of life | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30). Scores range fro 0 to 100, a higher score represents a higher (better) level of functioning or a higher (worse) level of symptoms.
Change in daily functioning and global quality of life | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30). Scores range fro 0 to 100, a higher score represents a higher (better) level of functioning or a higher (worse) level of symptoms.
Change in subjective well-being | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the Satisfaction with Life Scale. Total score range from 5 to 35, with increasing score implying higher subjective well-being.
Change in vitality | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the Subjective Vitality Scale. The total score ranges from 6 to 36 with a higher score indicating a better condition
Change in general health | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by European Quality of Life Five-dimension Scale Questionnaire (EQ-5D). Total score range from 5 (worst health) to 25 (best health).
Change in work ability | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by Work Ability Index. Total score range from 7 to 49 points, with higher score indicating better work ability.
Change in work ability | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by Work Ability Index. Total score range from 7 to 49 points, with higher score indicating better work ability.
Change in work ability | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by Work Ability Index. Total score range from 7 to 49 points, with higher score indicating better work ability.
Change in anxiety symptoms | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the General Anxiety Disorder 7-items. Total score range from 0 to 21 with increasing score implying higher level of anxiety.
Change in anxiety symptoms | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by the General Anxiety Disorder 7-items. Total score range from 0 to 21 with increasing score implying higher level of anxiety.
Change in anxiety symptoms | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by the General Anxiety Disorder 7-items. Total score range from 0 to 21 with increasing score implying higher level of anxiety.
Change in depressive symptoms | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the Patient Health Questionnaire-9. Total score from 0 to 27, increasing score implying higher depressive symptoms.
Change in depressive symptoms | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by the Patient Health Questionnaire-9. Total score from 0 to 27, increasing score implying higher depressive symptoms.
Change in depressive symptoms | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by the Patient Health Questionnaire-9. Total score from 0 to 27, increasing score implying higher depressive symptoms.
Change in level of physical activity | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the Godin Leisure Time Exercise Questionnaire
Change in level of physical activity | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by the Godin Leisure Time Exercise Questionnaire
Change in level of physical activity | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by the Godin Leisure Time Exercise Questionnaire
Change in exercise mastery | Change from baseline (week 0) and to post-intervention (week 13)
  Assessed by the Perceived Competence Scale. The scale consists of 4 items (statements). On each item, participants are asked to rate how true a statement is using a 7-point scale.Total score range from 4 to 28, with increasing score reflecting higher exercise mastery.
Change in exercise mastery | Change from baseline (week 0) to 4 months follow-up (week 29)
  Assessed by the Perceived Competence Scale. The scale consists of 4 items (statements). On each item, participants are asked to rate how true a statement is using a 7-point scale.Total score range from 4 to 28, with increasing score reflecting higher exercise mastery.
Change in exercise mastery | Change from baseline (week 0) to 7 months follow-up (week 42)
  Assessed by the Perceived Competence Scale. The scale consists of 4 items (statements). On each item, participants are asked to rate how true a statement is using a 7-point scale.Total score range from 4 to 28, with increasing score reflecting higher exercise mastery.
Change in dietary intake of the participants | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by a digital food frequency questionnaire (DIGIKOST-FFQ)
Change in meal pattern | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by the Meal Pattern Questionnaire
Change in body mass index | Change from baseline (week 0) and to post-intervention (week 13)
  Calculated by measuring weight and height
Change in body mass index | Change from baseline (week 0) to 4 months follow-up (week 29)
  Calculated by measuring weight and height
Change in body mass index | Change from baseline (week 0) to 7 months follow-up (week 42)
  Calculated by measuring weight and height
Change in sleep problems | Change from baseline (week 0) and to post-intervention (week 13)
  Measured by questions from the Trøndelag Health Survey
Change in sleep problems | Change from baseline (week 0) to 4 months follow-up (week 29)
  Measured by questions from the Trøndelag Health Survey
Change in sleep problems | Change from baseline (week 0) to 7 months follow-up (week 42)
  Measured by questions from the Trøndelag Health Survey
Change in cardiorespiratory fitness | Change from baseline (week 0) and to post-intervention (week 13)
  Assessed by a submaximal and indirect treadmill test (modified Balke protocol)
Change in cardiorespiratory fitness | Change from baseline (week 0) to 4 months follow-up (week 29)
  Assessed by a submaximal and indirect treadmill test (modified Balke protocol)
Change in cardiorespiratory fitness | Change from baseline (week 0) to 7 months follow-up (week 42)
  Assessed by a submaximal and indirect treadmill test (modified Balke protocol)
Change in lower body muscle strength | Change from baseline (week 0) and to post-intervention (week 13)
  Assessed by 30 second sit-to-stand test
Change in lower body muscle strength | Change from baseline (week 0) to 4 months follow-up (week 29)
  Assessed by 30 second sit-to-stand test
Change in lower body muscle strength | Change from baseline (week 0) to 7 months follow-up (week 42)
  Assessed by 30 second sit-to-stand test
Change in upper body muscle strength | Change from baseline (week 0) and to post-intervention (week 13)
  Assessed by maximum repetitions of push-ups with various starting positions
Change in upper body muscle strength | Change from baseline (week 0) to 4 months follow-up (week 29)
  Assessed by maximum repetitions of push-ups with various starting positions
Change in upper body muscle strength | Change from baseline (week 0) to 7 months follow-up (week 42)
  Assessed by maximum repetitions of push-ups with various starting positions
Change in quality of life among relatives | Change from baseline (week 0) and to post-intervention (week 13)
  Assessed by the Research and Development 36-item Short Form Survey (RAND SF-36).The eight scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better quality of life.
Change in global health status among relatives | Change from baseline (week 0) and to post-intervention (week 13)
  The global health status / quality of life scale from the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30). Scores range from 0 to 100, a higher score represents a higher (better) level of functioning or a higher (worse) level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Thorsen, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Bohn S, Oldervoll LM, Reinertsen KV, Seland M, Fossa A, Kiserud C, Skaali T, Nilsen TS, Blomhoff R, Henriksen HB, Lie HC, Berge T, Fjerstad E, Wisloff T, Slott M, Zajmovic I, Thorsen L. The feasibility of a multidimensional intervention in lymphoma survivors with chronic fatigue. Support Care Cancer. 2023 Dec 14;32(1):22. doi: 10.1007/s00520-023-08204-5. PMID 38095797